#### 1. TITLE PAGE

STUDY TITLE A Double-Blind, Randomized, Placebo-Controlled, Parallel

Group, Three-Arm, Multi-Site Study to Evaluate the Clinical Equivalence of Diclofenac Sodium Topical Gel 1% (Hi-Tech Pharmacal Co., Inc.) with Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis) in Patients with Osteoarthritis of the

Knee

SPONSOR Hi-Tech Pharmacal Co., Inc.

Address: 369 Bayview Avenue Amityville, NY, 11701, USA

PROTOCOL NUMBER OGD protocol #P130021 assigned by the FDA in its April 16,

2015 letter

STUDY Bioequivalence Study with Clinical Endpoint

CLASSIFICATION

INVESTIGATIONAL Test Product: Diclofenac Sodium Topical Gel 1% (Hi-Tech

PRODUCT Pharmacal Co., Inc.)

Reference Product: Voltaren® Gel (Diclofenac Sodium Topical

Gel) 1% (Novartis)

Placebo: Topical gel (vehicle) with no active ingredient

INDICATION Pain associated with osteoarthritis of knee

DOSE Subjects were randomized to receive a 4 gram dose of the generic

Diclofenac Sodium Topical Gel, 1% (Test), the Reference Listed Drug (RLD), or Placebo applied to the arthritic knee four times

daily for eight (8) weeks.

STUDY POPULATION All included subjects were at least 35 years of age, of either sex,

of any race, were diagnosed with osteoarthritis of the knee in one or both knees and met all inclusion criteria and none of the

exclusion criteria.

FIRST PATIENT December 8, 2014

TREATED

Version 2.0 1 | P a g e

Clinical Study Report DICL001

Hi-Tech Pharmacal Co., Inc. Confidential

LAST PATIENT April 01, 2016

COMPLETED

SPONSORS Biswajit Pati, Ph.D., Senior Vice President, Research &

RESPONSIBLE Development

MEDICAL OFFICER

SPONSOR Biswajit Pati, Ph.D., Senior Vice President, Research &

REPRESENTATIVE Development

Responsibility: Sr. VP, Research and Development

Akom Pharmaceuticals, Inc.

1925 West Field Court, Suite 300, Lake Forest, IL 60045, USA

Tel: 847-353-4966 Fax: 847-279-6191

Email: Biswajit.pati@akorn.com

DATE June 21st, 2018

This study was performed in accordance with Good Clinical Practice, the ethical principles that have their origin in the Declaration of Helsinki and the applicable regulatory agency requirements including Title 21 of the Code of Federal Regulations 50, 56, and 312, the EU Directives 2001/20/EC and 2005/28/EU, and the International Conference on Harmonization Guideline E6. The information in this document is confidential. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the sponsor.

Version 2.0 2 | P a g e

Hi-Tech Pharmacal Co., Inc. Confidential

#### 2. SYNOPSIS

NAME OF Hi-Tech Pharmacal Co., Inc.

SPONSOR/COMPANY

NAME OF FINISHED Diclofenac Sodium Topical Gel 1%

PRODUCT

NAME OF ACTIVE Diclofenae Sodium

INGREDIENT

STUDY TITLE A Double-Blind, Randomized, Placebo-Controlled, Parallel Group,

Three-Arm, Multi-Site Study to Evaluate the Clinical Equivalence of Diclofenac Sodium Topical Gel 1% (Hi-Tech Pharmacal Co., Inc.) With Voltaren® Gel (Diclofenac Sodium Topical Gel) 1%

(Novartis) in Patients with Osteoarthritis of the Knee

INVESTIGATORS The entire listing of all Investigators can be found in Appendices

16.1.4.1-16.1.4.6

STUDY CENTRES 55 centers in Ukraine, Poland, Romania, Lithuania, Latvia and

Estonia

STUDY PERIOD 8 December 2014 (first patient in for the first protocol version) to

01 April 2016 (last patient out)

PHASE OF Bioequivalence Study with Clinical Endpoint

DEVELOPMENT

OBJECTIVES The objectives of the study were to demonstrate efficacy and safety

of Hi-Tech Pharmacal Co., Inc's Diclofenac Sodium Topical Gel 1% compared to Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis) in the treatment of patients with osteoarthritis of the

knee.

DESIGN This study followed a double-blind, randomized, placebo-

controlled, parallel group, three-arm, multi-site, 5-treatment visit study design with 934 subjects. Study centers (in several European countries) participated in this study to achieve approximately 800 modified Intention-to-Treat (ITT) patients, in order to complete at least 750 Per Protocol (PP) patients. Patients were randomized

Version 2.0 3 | P a g e

1:1:1 to receive the Test Product, or the Reference Product, or Placebo treatment, respectively.

Patients with osteoarthritis (OA) of the knee were asked to administer the study medication four (4) times daily for eight (8) weeks. Patients visited the study site as per the following visit schedule:

Visit 0/Screening - Day -9±2

Visit 1/Baseline - Day 0

Visit 2/Week 2 - Day 14±2

Visit 3/Week 4 - Day 28±2

Visit 4/Week 6 - Day 42±2

Visit 5 - Day 56±2/Termination Visit

Visits were calculated based on Visit 1 Day 0. A window of ±2 days was allowed for each visit (other than Visit 1) however the total duration of study drug administration could not exceed 8 weeks ±2 days.

The initial protocol versions prior to the protocol version 1.9 had the following study schedule to accommodate the placebo run-in during the pain medication washout period (between Visits 0 and 1):

Visit -1/Prescreening - Day -30 to -10

Visit 0/Screening - Day -7

Visit 1/Baseline - Day 0

Visit 2/Week 2 - Day 14±2

Visit 3/Week 4 - Day 28±2

Visit 4/Week 6 - Day 42±2

Visit 5/Week 8 - Day 56±2

In its April 16, 2015 response to our protocol DICL001 (its initial version 1.5 was submitted to the FDA OGD on September 24, 2013), the OGD disagreed with our proposed use of placebo gel during the pain medication washout period and hence the protocol was modified accordingly.

Version 2.0

SAMPLE SIZE, Planned: 900 subjects in total with 300 subjects in each treatment

PLANNED AND group

ANALYZED Analyzed: 934 subjects in total with 316 subjects who received Test

Product, 312 Reference Product and 306 Placebo

Enrolled: 934 Screened: 1039

INDICATION Pain associated with osteoarthritis of knee

MAIN CRITERIA FOR 1. Ambulatory male and non-pregnant females 35 years and older

INCLUSION diagnosed with osteoarthritis according to the American College of (PROTOCOL Rheumatology Criteria (ACR) in one knee. Target knee is the one

VERSION 1.9)\* with higher level of pain.

ACR Criteria includes: Knee Pain and at least 3 of the following:

1) age  $\geq 50$ 

2) stiffness lasting < 30 mins

3) bony tenderness

4) crepitus

5) bony enlargement

6) no palpable warmth

Symptom onset of > 6 Months prior to Screening for the target knee.

- 3. If female and of child-bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., IUD, oral, transdermal, injected, implanted hormonal contraceptives or condom + spermicide).
- Periarticular knee pain due to osteoarthritis (not bursitis, tendonitis etc.) that required the use of oral or topical treatments (e.g., NSAIDs or acetaminophen).
- Radiograph of the target knee within the previous year with a Grade 1, 2 or 3 disease based upon the Kellgren-Lawrence disease severity scale.
- 6. After a minimum of 7-day wash out of all pain medication has

Version 2.0 5 | P a g e

#### Hi-Tech Pharmacal Co., Inc. Confidential

Baseline pain on movement score of  $\geq$  50mm on a 0-100-mm Visual Analogue Scale for the target knee.

- 7. After a minimum of 7-day wash out of all pain medication has Baseline WOMAC Pain sub scale of ≥ 9 on a 5 question, 5 point (0 to 4) Likert scale for the target knee.
- Willing and able to use only acetaminophen as rescue medication.
- 9. Willing and able to comply with the study requirements.

MAIN CRITERIA FOR EXCLUSION (PROTOCOL VERSION 1.9)\*

- Females who are pregnant, breast feeding, or planning a pregnancy.
- Radiograph of the target knee within the previous year with a Grade 4 score on the Kellgren-Lawrence disease severity scale.
- History of osteoarthritis in the contralateral knee requiring medication (OTC or prescription) within 12 months of screening.
- 4. After a minimum of 7-day wash out of all pain medication has Baseline pain on movement score of ≥ 20mm on a 0-100-mm Visual Analogue Scale for the contralateral knee immediately prior to randomization.
- Known history of secondary osteoarthritis (e.g. congenital, traumatic, gouty arthritis) of the knee or rheumatoid arthritis.
- 6. Known history of other chronic inflammatory diseases, (e.g., colitis) or fibromyalgia during last 5 years. Patients whose disease was diagnosed at least 5 (five) years prior to screening visit and have had no known disease activity (i.e., neither disease related complaints nor disease treatment prescribed) since then may enter in the study.
- 7. History of asthma, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease. Patients who have had high blood pressure measured at least 2 (two) years prior to screening visit and have had no disease activity (i.e., no record of hypertension or antihypertensive treatment prescribed) for at least 2 (two) years prior to

Version 2.0 6 | P a g e

screening visit may enter in the study.

- 8. History of coronary artery bypass graft within 6 months of screening.
- 9. Concomitant acetylsalicylic acid therapy other than a stable low dose used for cardiac prophylaxis (max. 162 mg daily) taken for at least 3 months prior to enrollment and maintained throughout the duration of the study.
- Use of warfarin or other anticoagulant therapy within 30 days of screening.
- Use of ACE inhibitors, cyclosporine, diuretics, lithium or methotrexate, within 30 days of screening or during the study.
- Known history of gastrointestinal bleeding or peptic ulcer disease.
- Abnormal screening clinical laboratory evaluations which the Investigator deems clinically significant.
- 14. Known allergy to aspirin or NSAIDs.
- 15. Skin lesions or wounds in the affected area.
- 16. Significant (requiring surgery) injury or major knee surgery to either knee within six months prior to screening.
- Transaminase levels that are more than two times the upper limit of the normal range at screening.
- 18. Any other acute or chronic illness that in the opinion of the investigator could compromise the integrity of study data or place the Patient at risk by participating in the study.
- Concomitant use of corticosteroids (any formulation) or use within 30 days of study randomization.
- 20. Receipt of any drug as part of a research study within 30 days prior to screening.
- 21. Previous randomization into this study.
- 22. Known allergy (hypersensitivity) to acetaminophen.
- \* the inclusion and exclusion criteria of the earlier protocol versions are in the DICL001 protocols file and Chapter 9.8 of this

Version 2.0 7 | P a g e

CSR.

TEST PRODUCT. In:

Investigational drug (Test Product): Diclofenac Sodium Topical Gel

DOSE AND MODE OF

1% (Hi-Tech Pharmacal Co., Inc.)

ADMINISTRATION

Dosage and regimen: Test Drug was used on knees to treat arthritis pain and was administered topically. Subjects applied 4 grams for 4

times a day (total dose for one day was 16 grams).

All subjects received medication from the following batches:

620576 (Diclofenac Sodium Topical Gel) W3633 or W4347 (Voltaren® Gel)

624354 (Placebo)

REFERENCE

Reference Product: Voltaren® Gel (Diclofenac Sodium Topical

PRODUCT: DOSE

Gel) 1% (Novartis)

AND MODE OF

Placebo: Topical gel (vehicle) with no active ingredient

ADMINISTRATION

Dosage and regimen: Reference Drug and Placebo were used on knees to treat arthritis pain and were administered topically. Subjects applied 4 grams four times a day (total dose for one day

was 16 grams).

All subjects received medication from the following batches:

620576 (Diclofenac Sodium Topical Gel) W3633 or W4347 (Voltaren® Gel)

624354 (Placebo)

DURATION OF

8 weeks ±2 days

STUDY FOR INDIVIDUAL SUBJECT

CRITERIA FOR

Criteria for Effectiveness:

EVALUATION

Bioequivalence for Test Drug is established if with 90% confidence the ratio of means of the WOMAC Pain scores for Test and RLD remains within 0.80 and 1.25. The sensitivity of the study will be acceptable if mean changes from Baseline in the WOMAC Pain scores for Test and RLD are statistically significantly greater (p<0.05) than that for the Placebo in the ANCOVA based on the Treatment and Placebo results.

### Safety Measures:

Safety measures will include the incidences of treatment emergent adverse events (reported, elicited and observed), abnormal vital signs, clinically significant changes from Baseline in physical examination results.

# STATISTICAL METHODS

#### For efficacy data:

- Descriptive evaluation of all endpoints
- Ratio of mean WOMAC Pain scores between Test and Reference Products and their 90% confidence interval.
- Parametric method (ANCOVA) for the comparison of Treatment versus Placebo in the mean change from Baseline in the WOMAC Pain score

### For safety evaluation:

Descriptive statistical methods

#### **ENDPOINTS**

# Primary Efficacy Endpoints

 Mean Change from Baseline to Week 8 in WOMAC Pain Scale

## Secondary Efficacy Endpoints

 Superiority of Test and Reference against Placebo in the Mean Change from Baseline to Week 8 in the total WOMAC Pain score.

### Safety Endpoints

- Incidences of treatment emergent adverse events
- Abnormal vital signs
- Clinically significant changes from Baseline in physical examination results.

Version 2.0 9 | P a g e